CLINICAL TRIAL: NCT02056847
Title: Randomized, Open-label, Multi-centered Study to Evaluate the Safety and Efficacy of Pitavastatin in Patients With Impaired Fasting Glucose and Hyperlipidemia(Phase 4)
Brief Title: to Evaluate the Safety and Efficacy of Pitavastatin in Patients With IFG and Hyperlipidemia
Acronym: SIPHON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Collaborators: The Catholic University of Korea (Other); Kyunghee University Medical Center (Other); Korea University Guro Hospital (Other); Dong-A University Hospital (Other); Seoul National University Bundang Hospital (Other); Samsung Medical Center (Other); Seoul National University Hospital (Other); Ajou University School of Medicine (Other); Gangnam Severance Hospital (Other); Severance Hospital (Other); Yeungnam University Hospital (Other); Ulsan University Hospital (Other); Eulji University Hospital (Other); Asan Medical Center (Other); Chonnam National University Hospital (Other); Chonbuk National University Hospital (Other); Chungnam National University Hospital (Other); Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JW-PTV-713
Record Dates: First submitted 2014-02-04; First posted 2014-02-06 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2017-03

CONDITIONS: HbA1c Level Associated With Lipid Compositions
Keywords: Livalo, pitavastatin, hyperlipidemia, IFG
MeSH Terms: conditions — Hyperlipidemias | interventions — pitavastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pitavastatin calcium 4mg (Active Comparator): Pitavastatin calcium (LIVALO®) 4mg, once a day
  Interventions: Drug: Pitavastatin calcium 4mg
- Pitavastatin calcium 2mg (Active Comparator): Pitavastatin calcium (LIVALO®) 2mg, once a day
  Interventions: Drug: Pitavastatin calcium 2mg

INTERVENTIONS:
Drug: Pitavastatin calcium 4mg — taking once a day
  Other Names: Pitavastatin calcium(LIVALO) 4mg
  Arms: Pitavastatin calcium 4mg
Drug: Pitavastatin calcium 2mg — Taking once a day
  Other Names: LIVALO 2mg
  Arms: Pitavastatin calcium 2mg

SUMMARY:
Primary Objective

: To evaluate that there is no different effect on HbA1c between routine lipid lowering therapy(Livalo 2mg) and intensive lipid lowering therapy(Livalo 4mg) in the hyperlipidemic patients with impaired fasting glucose (IFG).

H0: µT-µC ≥ 0.4 vs H1: µT-µC < 0.4

µT = the change of HbA1c in the test drug (Pitavastatin 4 MG) µC = the change of HbA1c in the control drug (Pitavastatin 2 MG)

DETAILED DESCRIPTION:
Investigational Product Test group: Pitavastatin calcium (LIVALO) 4mg tab Control group: Pitavastatin calcium (LIVALO) 2mg tab

Study Site: Multi-centers in Korea

Period: For 24months after IRB approval at each site (Including 12months of subject enrollment period)

Efficacy End points

A. Primary end point The change of HbA1c before and after taking LIVALO

B. Secondary end point

1. Incidence of diabetes within 1year after registration (based; FPG ≥126mg/dL or to need taking diabetes medication)
2. Incidence of major cardiovascular (TLR-MACE) events within 1 year after registration
3. Incidence of total cardiovascular (TVR-MACE) events within 1 year after registration
4. The change of the lipid composition (T-chol, TG, LDL-C, HDL-C, ApoA1/ApoB)
5. The changes of hs-CRP
6. The changes of Adiponectin
7. The change of blood glucose and Insulin levels FPG(Fasting Plasma Glucose) Fasting Serum Insulin HOMA IR [fasting insulin(µIU/mL) X fasting glucose(mg/dL)]/405 HOMA β [360 X fasting insulin(µIU/mL)]/[fasting glucose(mg/dL)-63]

Statistical Methods

1. Efficacy A. Primary efficacy endpoint analysis Describe statistics of basic about the HbA1c variation before and after taking LIVALO by groups. In order to verify noninferiority of test drug, check that upper limit of confidence interval of the one-sided 97.5% is less than 0.4% about difference of HbA1c variation between the control group and the test group, before and after taking LIVALO.

   B. Secondary efficacy endpoint analysis Continuous variables

   :Present the mean, standard deviation, minimum, and maximum values for TC, TG, LDL-C, HDL-C, Fasting serum insulin, Fasting plasma glucose and HOMA IR, HOMA β etc. by each visit and in each group. In comparison with intergroup, using two-sample t-test for normal distribution and using Wilcoxon rank sum test for non-normal distribution. Also In comparison with the same group, using paired t-test for normal distribution and using Wilcoxon signed rank test for non-normal distribution.

   Discrete variables

   : The number and percentage of the subjects for incidence of DM and cardiovascular event are described of each group and the ratio of the intergroup comparison use χ2-test or Fisher's exact test.
2. Safety All the AEs and the ADRs which manifested more than once are described by the frequency and percentage of each group and use χ2-test or Fisher's exact test for intergroup comparison about the rate of AEs and ADRs Laboratory tests and vital signs are analyzed descriptive statistics quantity of each group, and in comparison with intergroup, use two-sample t-test for normal distribution and use Wilcoxon rank sum test for non-normal distribution. Also, In comparison with the same group, use paired t-test for normal distribution and use Wilcoxon signed rank test for non-normal distribution.

Clinical laboratory test is analyzed the frequency and percentage of the outside normal range of subjects, and using χ2-test or Fisher's exact test with intergroup.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients who are more than 20 years old or 70 years old or less.
2. Patient who voluntarily sign on written informed consent form
3. Patient who LDL-C ≥ 100mg/dl or was diagnosed with hyperlipidemia
4. Patient who was suspected with Imparied Fasting Glucose (IFG) and satisfy FPG level ≥ 100mg/dL and < 126mg/dL when FPG measured twice.

Exclusion Criteria:

1. Patient who has familial hypercholesterolemia
2. Patient who has been diagnosed with Type1, Type2 DM or secondary DM(diabetes mellitus) at the screening visit (Diagnostic criteria of DM: HbA1c≥ 6.5%)
3. Patient who has received antidiabetic within 6weeks to the screening visit
4. Patient who has been taking insulin continuously or to be needed in the future
5. Patient who has a history of gastrectomy
6. Patient who is suspected or diagnosed with malignant tumor within last 10 years
7. Patient who has serious pancreatic disease or endocrine disorders
8. Patient who currently takes Cyclosporine
9. Patient who has a medical history of hypersensitivity to Pitavastatin calcium
10. Patient who has suspected renal failure (serum creatinine ≥2.0 mg/dL)
11. Patient who has suspected liver dysfunction (more than 2.5 times the upper limit of normal AST or ALT)
12. Patient who has more than 3 times the upper limit of normal CPK
13. Patient who is breastfeeding, pregnant or planning pregnancy
14. Patient who deemed inappropriate as subject in the opinion of the Principal Investigator or Investigator

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The change of HbA1c before and after taking LIVALO® | 24 weeks after taking IP

SECONDARY OUTCOMES:
Incidence of diabetes | within 1year after registration
  based; FPG ≥126mg/dL or to need taking diabetes medication
Incidence of total cardiovascular (TVR-MACE) events | within 1 year after registration
The change of the lipid composition (T-chol, TG, LDL-C, HDL-C, ApoA1/ApoB) | 24weeks and 1 year after registration
The changes of hs-CRP, Adiponectin, blood glucose and Insulin levels | 24weeks and 1 year after registration
  The change of blood glucose and Insulin levels FPG(Fasting Plasma Glucose) Fasting Serum Insulin HOMA IR [fasting insulin(µIU/mL) X fasting glucose(mg/dL)]/405 HOMA β [360 X fasting insulin(µIU/mL)]/[fasting glucose(mg/dL)-63]

CONTACTS AND LOCATIONS:
Overall Officials: NamSik Chung, M.D., Ph D., Principal Investigator — Severance Hospital
Locations (1):
- JW pharmaceutical, Seoul, South Korea